CLINICAL TRIAL: NCT03507283
Title: Outcomes of Vertical Split Conjunctival Autograft Using Fibrin Glue in Treatment of Primary Double-head Pterygia
Brief Title: Vertical Split Conjunctival Autograft in Double-head Pterygia
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, lecturer of ophthalmology, Benha University
Other Study IDs: benha19991
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Pterygium of Conjunctiva and Cornea
Keywords: Pterygium; double-headed; vertical
MeSH Terms: conditions — Pterygium Of Conjunctiva And Cornea; Pterygium | interventions — Wound Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Double head pterygia excision and repair — Complete excision of the pterygia was done. A free conjunctival autograft was obtained. The graft was divided vertically into two parts then secured into conjunctival defects.

SUMMARY:
15 eyes of 15 patients with primary double-headed pterygia that underwent vertical split conjunctival autograft pterygium surgery were retrospectively reviewed. All patients had primary double-headed pterygia. Recurrence was defined as fibrovascular proliferation over the limbus onto the cornea.

Vertical split conjunctival autograft using fibrin glue is an effective technique with good cosmetic results and low to no recurrence for primary double head pterygia treatment.

DETAILED DESCRIPTION:
The pterygium body was dissected from the sclera. Complete excision of the pterygium, subconjunctival Tenon's tissue and surrounding fibrovascular tissues followed.The conjunctival edge was trimmed. The corneal surface was gently scraped with a scalpel. The Same procedure was done on temporal pterygia. A free conjunctival autograft was obtained. The graft was divided vertically into two parts. The nasal part of the graft was cut from limbal attachment including limbal tissue; temporal part was left attached. The nasal part of the graft was moved to the nasal conjunctival defect and attached to the sclera with fibrin sealant (Tisseel; Baxter, Vienna, Austria). The Same procedure was done with the temporal part of the graft. The orientation of graft was ensured before securing it.

ELIGIBILITY:
Inclusion Criteria:

* Primary double-headed pterygia

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 15 eyes of 15 patients. The mean age of all patients was 36.92 ± 10.8 years. There were 9 males (60%) and 6 females (40%).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The recurrence rate | 1 year
  ﬁbrovascular tissue invading the cornea and expressed as a percentage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elhamaky TR, Elbarky AM. Outcomes of Vertical Split Conjunctival Autograft Using Fibrin Glue in Treatment of Primary Double-Headed Pterygia. J Ophthalmol. 2018 Dec 20;2018:9341846. doi: 10.1155/2018/9341846. eCollection 2018. PMID 30671262